CLINICAL TRIAL: NCT03279003
Title: Study of the Efficacy and Tolerance of Light Therapy by Light-emitting Diode (LED) in Sensitive Skin
Brief Title: Study of the Efficacy and Tolerance of Light Therapy in Sensitive Skin
Acronym: SENSILED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SENSILED (29BRC16.0179)
Record Dates: First submitted 2017-09-01; First posted 2017-09-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2021-12

CONDITIONS: Sensitive Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Light-emitting diode therapy (Experimental): Exposure to LED light
  Interventions: Device: LED light

INTERVENTIONS:
Device: LED light — An exposure to LED light will be carried out twice a week until improvement, maximum 8 weeks.

SUMMARY:
Light-emitting diode (LED) light therapy is increasingly used successfully and without adverse effects in diabetic leg ulcer, chronic low back pain, chronic myofacial pain in the neck and in several dermatoses such as acne, Psoriasis, alopecia areata and skin rejuvenation. A Korean study conducted in 2013 suggested its effectiveness in patients with sensitive skin in connection with rosacea, acne, eczema. The objective of the study is to perform a study in subjects with a sensitive skin without associated dermatosis.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the efficacy of light-emitting diode therapy in subjects with sensitive skin and to assess pain improvement, evaluation of improvement in pruritus and evaluation of treatment tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Age less than or equal to 70
* Sensitive skin defined by a score ≥ 40 on the Sensiscale scale
* Patient able to consent

Exclusion Criteria:

* Persons under 18 years of age or over.
* Persons suffering from disorders of higher functions preventing comprehension of the questionnaire.
* Pregnancy.
* Analgesic or medication acting on the nervous system.
* Other dermatosis of the face (example: rosacea, seborrheic dermatitis, acne ...).
* Neurological or psychiatric illness.
* A photosensitizing drug.
* Refusal of patient
* Patients under legal protection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of light therapy | 2 months
  The improvement of sensitive skin symptoms will be measured by the Sensiscale scale

SECONDARY OUTCOMES:
Assessment of pain improvement | 2 months
  Pain improvement will be done by self-evaluation of the patients, using a visual analog scale
Assessment of improvement in pruritus | 2 months
  The improvement of pruritus will be done by self-evaluation of the patients, using a visual analog scale
Assessment of the tolerance | 2 months
  At the end of the study, patients will be questioned about the possible occurrence of side effects listed in the patient's notebook during the 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

REFERENCES:
- [Result] Sonbol H, Brenaut E, Nowak E, Misery L. Efficacy and Tolerability of Phototherapy With Light-Emitting Diodes for Sensitive Skin: A Pilot Study. Front Med (Lausanne). 2020 Feb 7;7:35. doi: 10.3389/fmed.2020.00035. eCollection 2020. PMID 32118019